CLINICAL TRIAL: NCT00733473
Title: Phase 4 Study of Nebulized Budesonide for Children Who Are Hospitalized for Acute Wheezing
Brief Title: Nebulized Budesonide for Children Who Are Hospitalized for Acute Wheezing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kecioren Education and Training Hospital (Other)
Responsible Party: Principal Investigator, Cem Hasan Razi, MD, Kecioren Education and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B.10.0.İEG.0.11.00.01-3246
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Asthma; Acute Asthma
Keywords: Wheezing; Acute asthma; Children
MeSH Terms: conditions — Asthma; Respiratory Sounds | interventions — Budesonide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Budesonide (Active Comparator): This arm consist 50 children with recurrent wheezing who are hospitalized for wheezing epizode. They received 1 mg nebulized budesonide 2 times a day upto 5 days
  Interventions: Drug: Budesonide 0.5 mg/ml nebules
- 2 Placebo saline (Placebo Comparator): This arm consist 50 children with recurrent wheezing who are hospitalized for wheezing epizode. They received 2ml of nebulized saline 2 times a day upto 5 days
  Interventions: Drug: % 0.9 Saline solution

INTERVENTIONS:
Drug: Budesonide 0.5 mg/ml nebules — Children will receive 1 mg nebulized budesonide 2 times a day up to 5 days
  Other Names: Pulmicort 0.5 mg/ml nebules
  Arms: 1 Budesonide
Drug: % 0.9 Saline solution — Children will receive 2 ml of nebulized saline 2 times a day up to 5 days
  Arms: 2 Placebo saline

SUMMARY:
The purpose of this study is to determine if adding nebulized budesonide to the systemic steroid for treatment of acute wheezing has any additive benefit in children who have hospitalized for acute wheezing.

DETAILED DESCRIPTION:
Context: Inhaled steroids reduced admission rates in patients with acute asthma, but it is unclear if there is a benefit of inhaled corticosteroids when used in addition to systemic corticosteroids. There is insufficient evidence that inhaled corticosteroids result in clinically important changes in pulmonary function or clinical scores when used in acute asthma. Similarly, it was mentioned in the Cochrane Database of Systematic Reviews that further research is needed to clarify if there is a benefit of inhaled corticosteroids when used in addition to systemic steroids.

Objective: To determine if adding nebulized budesonide to the systemic steroid for treatment of acute wheezing in hospitalized children has any benefit on, symptom score, duration of hospitalization and time to discharge from hospital.

Study Design/Setting/Participants: A double-blind, randomized, controlled trial of nebulized budesonide versus placebo for children 6 months to 6 years of age who have admitted to the hospital for acute wheezing.

Intervention: Participants will receive standard therapy including SCS, albuterol, and ipratropium bromide and will be randomly assigned to also receive either nebulized BIS or saline.

Study Measures: Differences in asthma scores, vital signs, duration of hospitalization and time to discharge from hospital will be compared between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Children who have recurrent wheezing attacks
* Children who admitted to the hospital for acute wheezing
* Clinical asthma score of 3-9
* Parental/guardian permission (informed consent) and if appropriate, child assent

Exclusion Criteria:

* Systemic corticosteroid use in the last 30 days
* Chronic lung diseases including cystic fibrosis
* Immunodeficiency
* Cardiac disease requiring surgery or medications
* Adverse drug reaction or allergy to budesonide, albuterol, ipratropium bromide, prednisone, prednisolone, or methylprednisolone
* Known renal or hepatic dysfunction
* Impending respiratory failure requiring positive pressure ventilation
* Immune deficiency
* Gastroesophageal reflux disease
* Suspected foreign body aspiration or croup
* Anatomic abnormalities of the respiratory tract

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Time to discharge from the hospital to home | 1-5 days

SECONDARY OUTCOMES:
Pulmonary index score | 1 to 5 days
Respiratory rate | 1 to 5 days
Oxygen saturation | 1 to 5 days
Adverse reactions. | 1 to 5 days

CONTACTS AND LOCATIONS:
Overall Officials: C H Razi, MD, Study Director — Kecioren Education and Training Hospital; C H Razi, MD, Principal Investigator — Kecioren Education and Training Hospital
Locations (1):
- Kecioren Education and Training Hospital, Ankara, Kecioren, Turkey (Türkiye)